CLINICAL TRIAL: NCT04106518
Title: Study of Genetic Determinants in Alcoholic Hepatitis and Establishment of a Multicenter Prospective Cohort of Patients With Alcoholic Liver Disease
Acronym: COMADHAA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2017_51; 2018-A02286-49 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2019-06-27; First posted 2019-09-27 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Alcoholic Liver Disease; Severe Alcoholic Hepatitis; Alcoholic Cirrhosis
Keywords: Cohort; alcoholic hepatitis; alcoholic cirrhosis; pathophysiology; bio bank; pan-genomic study
MeSH Terms: conditions — Liver Diseases, Alcoholic; Hepatitis, Alcoholic; Liver Cirrhosis, Alcoholic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — serum, plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- cirrhosis: Patients with alcoholic liver disease without alcoholic hepatitis
- severe alcoholic hepatitis: Patients with severe alcoholic hepatitis ( Maddrey score ≥32)
- non-severe alcoholic hepatitis: Patients with non-severe alcoholic hepatitis (Maddrey score <32)

SUMMARY:
Alcoholic hepatitis carries a risk of high mortality at short term, especially in its severe form. Its diagnosis is confirmed by liver biopsy. The prevalence of alcoholic hepatitis, severe or not severe, is poorly known and prospective data are needed. The present observational study aims to define the prevalence of alcoholic hepatitis among patients admitted for jaundice and determine their outcome according to the severity. Survival and markers of liver dysfunction will be assessed. A biobank including genetic samples will be created to identify the disease profile in terms of inflammation and regeneration. The performance of non-invasive criteria for diagnosis will also be studied.

ELIGIBILITY:
Inclusion Criteria:

For SAH group:

* Alcohol consumption :

  * On average> 40 g / day for women and 50 g / day for men
  * Duration:> 5 years
* Recent jaundice episode (less than 3 months)
* Bilirubin> 50 mg / l (85μmol / l)

For NSAH group:

- Alcohol consumption :

* On average> 40 g / day for women and 50 g / day for men
* Duration:> 5 years

For cirrhosis (control) group:

* Alcohol consumption :

  * On average> 40 g / day for women and 50 g / day for men
  * Duration:> 5 years
* Unambiguous presence of cirrhosis criteria, including:

  * clinical signs (ascites, stellar angiomas ...) and / or
  * radiological signs (scanner or MRI: signs of hepatic dysmorphism and / or portal hypertension) and / or
  * biological signs (increased INR, thrombocytopenia) and / or
  * endoscopic signs (oesophageal / gastric varices)

Exclusion Criteria:

For NAH and NSAH groups:

* Presence of another hepatic pathology: evidenced by blood biology, imaging or histology (viral or autoimmune hepatitis, hemochromatosis, Wilson's disease)
* Presence of hepatocellular carcinoma
* HIV infection

For cirrhosis (control) group:

* History established / suggestive of HAA (Clinical, biological and / or histological criteria) in particular absence of jaundice episode
* Presence of another hepatic pathology: evidenced by blood biology, imaging or histology (viral or autoimmune hepatitis, hemochromatosis, Wilson's disease)
* Presence of hepatocellular carcinoma
* HIV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to jaundice will receive a liver biopsy in accordance with the usual management for diagnosis of alcoholic hepatitis, according to the recommendations of the European Association of Liver Diseases (EASL).
Sampling Method: Probability Sample
Enrollment: 447 (Estimated)
Dates: Start 2019-10-23 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Prevalence of alcoholic hepatitis in heavy drinkers with jaundice | At baseline (time of liver biopsy)
  Assess the prevalence of biopsy-proven alcoholic hepatitis in a cohort of heavy drinkers admitted with recent jaundice

SECONDARY OUTCOMES:
Survival | at 12 months
  Survival rate at 12 months
Change in serum total bilirubin | Baseline, at 7 days, at 30 days, at 3 months at 6 months and at 12 months
  Total bilirubin is a liver parameter, used for the biological liver test evaluation, measured in mg/dl in the serum
Change in serum creatinine | Baseline, at 7 days, at 30 days, at 3 months at 6 months and at 12 months
  Creatinine is a marker of kidney function, assessed in the blood and measured in milligrams per deciliter
Change in MELD (Model for End-stage Liver Disease)score | Baseline, at 7 days, at 30 days, at 3 months at 6 months and at 12 months
  The MELD score is a validated tool based on INR, creatinine and bilirubin measured in the blood with the following formula:(9.57 × log creatinine in milligrams per deciliter) + (3.78 × log bilirubin in milligrams per deciliter) + (11.20 × log international normalized ratio) + 6.43. The MELD score is used in liver disorders to assess the degree of liver failure. It has no unit.
Identification of inflammatory and biochemical profiles of patients with severe, non-severe and cirrhotic alcoholic hepatitis, based on the constitution of a biobank (serum and plasma) | Baseline, at 7 days, at 30 days and at 12 months
  Serum and plasma evaluation of translational markers (e.g. cytokines) associated with inflammation in patients with alcohol-related liver disease. The list of markers which will be assessed cannot be determined at present and will depend on other ongoing studies performed in alcoholic hepatitis.
Identification of the genetic profiles of individuals with severe, non-severe and cirrhotic alcoholic hepatitis( blood sample) | Baseline
  Evaluation of genetic markers associated with alcoholic hepatitis as compared to patients with alcohol-related liver disease without alcoholic hepatitis. We will use a non a priori approach as recommended in genetic studies. Thus, the list of genetic markers cannot be provided at that time.
Measurement of diagnostic performance (area under the ROC curve) | At baseline
  Measurement of diagnostic performance (area under the ROC curve) of the simple and non-invasive clinical and biological criteria for alcoholic hepatitis proposed in an international expert opinion

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Louvet, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (9):
- France (9):
  - Chr Angers, Angers
  - Chru Besancon, Besançon
  - Hôpital Jean Verdier, AH-HP, Bondy
  - Centre Hospitalier Universitaire, Caen
  - Hopital Nord - Chu38 - La Tronche, La Tronche
  - Hôpital Claude Huriez, CHU, Lille
  - Association Hopital Saint Joseph - Marseille, Marseille
  - Chu Montpellier, Montpellier
  - Hu Est Parisien Site St Antoine Aphp - Paris 12, Paris